CLINICAL TRIAL: NCT02663141
Title: Randomized Clinical Trial of Intravitreal Bevacizumab Versus Intravitreal Bevacizumab Combined With Losartan in the Treatment of Diabetic Macular Edema
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Collaborators: Farabi Eye Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9111257006
Record Dates: First submitted 2016-01-21; First posted 2016-01-26 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — Losartan; Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Losartan (Experimental): Oral losartan 50 mg daily for 6 months
  Interventions: Drug: Losartan; Drug: Intravitreal bevacizumab
- Placebo (Placebo Comparator): Oral placebo daily for 6 months
  Interventions: Drug: Intravitreal bevacizumab; Drug: Placebo

INTERVENTIONS:
Drug: Losartan
  Arms: Losartan
Drug: Intravitreal bevacizumab
  Other Names: Avastin
Drug: Placebo
  Arms: Placebo

SUMMARY:
The aim of this study is to determine whether oral losartan is effective in the treatment of diabetic macular edema (DME) as an adjuvant for intravitreal bevacizumab (IVB).

ELIGIBILITY:
Inclusion Criteria:

All type 2 diabetes mellitus patients with clinically significant macular edema(CSME), except those mentioned as exclusion criteria

Exclusion Criteria:

1. Patients with Uncontrolled hypertension
2. Patients with Proliferative diabetic retinopathy
3. Patients Who received angiotensin converting enzyme inhibitor(ACEI) or angiotensin receptor blocker(ARB)
4. Previous treatment for diabetic retinopathy (e.g., laser photocoagulation, photodynamic therapy, intravitreal injections of steroids, or anti-vascular endothelial growth factor, retinal surgery)
5. media opacities
6. evidence of any other ocular disease(e.g., glaucoma, uveitis, age related macular degeneration or etc.,)
7. Pathologic myopia > 6 Diopter
8. Patients with poor fixation or cooperation
9. Patients with renal or cardiac disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2015-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
difference in ETDRS best-corrected visual acuity (BCVA) between arms | Within 6 months from therapy
Difference in frequency of intravitreal Bevacizumab injection between arms | Within 6 months from therapy

SECONDARY OUTCOMES:
change in central macular thickness(measured by spectral domain optical coherence tomography) | Within 6 months from therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Farabi Eye Hospital, Tehran, Tehran Province, Iran